CLINICAL TRIAL: NCT06928714
Title: Pediatric Feeding Disorder Evolution in Amiens University Hospital
Acronym: EVOLTOA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2025_843_0019
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Feeding Disorders; Eating Behaviors; Dysphagia; Nutritional Status; Malnutrition; Children
Keywords: feeding disorders; eating behavior; dysphagia; nutritional status; malnutrition; artificial nutrition; children
MeSH Terms: conditions — Feeding and Eating Disorders; Feeding Behavior; Deglutition Disorders; Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Pediatric feeding disorders (PFDss) affect children with age-inappropriate oral intakes lasting at least 2 weeks, associated with medical, nutritional, psychosocial or feeding skills dysfunction. Feeding is a complex function involving the digestive tract, and different structures. It evolves throughout the child's development. It involves the caregiver-child relationship. Dysfunction of one or more of these systems may be the cause of pediatric feeding disorders. PFDs affect 25% of children, 5% with severe forms. PFDs can have severe nutritional consequences. They often cause malnutrition, even undernutrition, and sometimes overweight.

ELIGIBILITY:
Inclusion Criteria:

* Children <18 years old
* with at least two pediatric gastroenterology PFDs consultations at CHUAP ,
* with an inapropriate oral intakes for at least 2 weeks,
* Association with medical, nutritional, psychosocial or eating-skills dysfunction.

Exclusion Criteria:

* anorexia nervosa

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children <18 years old with at least two pediatric gastroenterology PFDs consultations at CHUAP , with an inapropriate oral intakes for at least 2 weeks, Association with medical, nutritional, psychosocial or eating-skills dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of children with Pediatric feeding disorders disappearance | 6 months
  Frequency of children with Pediatric feeding disorders disappearance

SECONDARY OUTCOMES:
Frequency of children with Pediatric feeding disorders disappearance | 1 year
Frequency of children with Pediatric feeding disorders disappearance | 2 years
Frequency of children with Pediatric feeding disorders disappearance | 3 years
Frequency of children with Pediatric feeding disorders disappearance | 5 years
Frequency of children with Pediatric feeding disorders disappearance | 8 years
Frequency of children with Pediatric feeding disorders disappearance | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No